CLINICAL TRIAL: NCT04702295
Title: COVID Vaccination in Rare and Complex Connective Tissue Diseases: ERN ReCONNET Multicentre Prospective Cohort Study
Brief Title: ERN ReCONNET Study on COVID-19 Vaccination in Rare and Complex Connective Tissue Disease (VACCINATE)
Acronym: VACCINATE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Marta Mosca, Full Professor in Rheumatology, University of Pisa
Other Study IDs: UPISA2
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Connective Tissue Diseases; Rare Diseases; Rheumatologic Disorder
MeSH Terms: conditions — Connective Tissue Diseases; Rare Diseases; Collagen Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
30 months, multicentre, prospective observational study on adult (>18 years) patients with a diagnosis of rare and complex connective tissue diseases (rCTDs) who will be given the vaccine during the period from January 2021 and January 2022.

Patients with the following diagnosis will be included:

* antiphospholipid syndrome (APS),
* Ehlers-Danlos syndrome (EDS),
* idiopathic inflammatory myopathies (IIM),
* IgG4-related disease (IgG4),
* mixed connective tissue disease (MCTD),
* relapsing polychondritis (RP),
* Sjogren's syndrome (SS),
* systemic lupus erythematosus (SLE),
* systemic sclerosis (SSc)
* undifferentiated connective tissue disease (UCTD)

DETAILED DESCRIPTION:
This is an observational study aimed at gathering sufficient number of cases of rCTDs patients who will receive COVID-19 vaccination that will help in better understanding of both safety and efficacy of the vaccine in this population. The study will be promoted both in ERN ReCONNET Full Members and Affiliated Partners as well as in other centres treating and managing rare and complex connective tissue diseases.

Study Objectives

1. To promote a harmonised data collection approach on COVID-19 vaccination in rare and complex CTDs patients;
2. To evaluate the safety profile of COVID-19 vaccination in rCTDs patients and to highlight possible disease-specific adverse events;
3. To evaluate the efficacy of COVID-19 vaccination in rCTDs patients and to highlight potential variables that prevent an effective immunization against COVID-19;
4. To evaluate differences in term of efficacy and safety among different types of vaccines in rCTDs patients
5. To depict the ideal patient's profile that would mostly benefit from COVID-19 vaccination

ELIGIBILITY:
Inclusion Criteria:

Patients with the following diagnosis will be included:

* antiphospholipid syndrome (APS),
* Ehlers-Danlos syndrome (EDS),
* idiopathic inflammatory myopathies (IIM),
* IgG4-related disease (IgG4),
* mixed connective tissue disease (MCTD),
* relapsing polychondritis (RP),
* Sjogren's syndrome (SS),
* systemic lupus erythematosus (SLE),
* systemic sclerosis (SSc)
* undifferentiated connective tissue disease (UCTD)

Exclusion Criteria:

* Pregnancy
* All the exclusion criteria that apply for COVID-19 vaccination in the general population

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult (>18 years) patients with a diagnosis of rCTDs who will be given the vaccine during the period from January 2021 and January 2022.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (any type) | 12 months
COVID-19 incidence in patients with and without evidence of past SARS-CoV-2 infection before and during vaccination regimen - cases confirmed ≥7 days after the last dose | 12 months

SECONDARY OUTCOMES:
Incidence of disease flare post-vaccination | 12 months
Incidence of serious adverse events | 12 months
Incidence of life-threatening adverse events and deaths | 12 months
Incidence of adverse events of special interest for COVID-19 | 12 months
Clinical variables (age, sex, underlying disease, ongoing treatment, comorbidities) associated with COVID-19 occurrence during the post-vaccination follow-up | 12 months
Comparison of the incidence of COVID-19 among different types of vaccines | 12 months
Significant anti COVID 19 antibodies titer at 3 and 6 months | 3 and 6 months